CLINICAL TRIAL: NCT04718922
Title: Effect of Chlorhexidine Mouthrinse on Prevention of Microbial Contamination During EBUS-TBNA: a Randomized Clinical Trial
Brief Title: Chlorhexidine Mouthrinse Before EBUS-TBNA
Acronym: CHX_EBUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeyoung Cho, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20110961173
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Endobronchial Ultrasound
Keywords: Endobronchial ultrasound; Transbronchial needle aspiration; Chlorhexidine; Infection; Complication
MeSH Terms: conditions — Infections | interventions — chlorhexidine gluconate; Mouthwashes

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Mouthrinse with 100 ml 0.12% chlorhexidine for 1 min
  Interventions: Drug: Chlorhexidine Gluconate 0.12 % Mouthwash
- Control Arm (No Intervention): No mouthrinse

INTERVENTIONS:
Drug: Chlorhexidine Gluconate 0.12 % Mouthwash — Intervention with chlorhexidine mouthrinse will be performed approximately 10 min before the start of EBUS-TBNA
  Other Names: Hexamedine Sol.
  Arms: Experimental Arm

SUMMARY:
The purpose of this study is to investigate whether chlorhexidine mouthrinse is effective in preventing microbial contamination during endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA).

DETAILED DESCRIPTION:
EBUS-TBNA using the convex probe is a standard of care for the assessment of mediastinal and hilar lymphadenopathy. Although EBUS-TBNA is a minimally invasive procedure, rare but serious infectious complications such as pneumonia, lung abscess, empyema, mediastinal adenitis/abscess, mediastinitis, pericarditis, and sepsis were reported. EBUS-scope might be contaminated with oropharyngeal commensal bacteria while passing the oropharyngeal airway during EBUS-TBNA. Contamination of punctured lymph nodes by oropharyngeal commensal bacteria can cause severe infections.

Chlorhexidine gluconate is an antimicrobial agent that has a broad antibacterial activity including both gram-positive and negative bacteria. Chlorhexidine has been widely used for surgical scrub, skin disinfection, and mouthrinse. We, therefore, designed a phase 4, single-center, randomized, controlled clinical trial to investigate whether chlorhexidine mouthrinse is effective in preventing microbial contamination during EBUS-TBNA.

ELIGIBILITY:
Inclusion Criteria:

* inpatients aged 19 years and older who are scheduled to undergo EBUS-TBNA using a convex probe

Exclusion Criteria:

* antiseptic mouthrinse within 7 days before inclusion;
* active infection or antibiotic treatment within 7 days before inclusion;
* immunocompromised;
* trachemostomy status;
* who have already undergone gastroscopy on the same day when EBUS- TBNA is scheduled to be administered

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Colony forming unit (CFU) counts of EBUS-TBNA needle wash solution in aerobic media | Needle wash solution is obtained immediately after termination of EBUS-TBNA
  Needle wash solution is obtained by instilling 5mL of sterile physiological saline into the puncture needle.

SECONDARY OUTCOMES:
CFU counts of EBUS-TBNA needle wash solution in anaerobic media | Needle wash solution is obtained immediately after termination of EBUS-TBNA
  Needle wash solution is obtained by instilling 5mL of sterile physiological saline into the puncture needle.
Fever | 24 hours after EBUS-TBNA
  Fever is defined as a temperature ≥37.8°C.
Infectious complications | 4 weeks after EBUS-TBNA
  Infectious complications include pneumonia, lung abscess, empyema, mediastinal adenitis/abscess, mediastinitis, pericarditis, and sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim NY, Park JH, Park J, Kwak N, Choi SM, Park YS, Lee CH, Cho J. Effect of chlorhexidine Mouthrinse on prevention of microbial contamination during EBUS-TBNA: a randomized controlled trial. BMC Cancer. 2022 Dec 20;22(1):1334. doi: 10.1186/s12885-022-10442-5. PMID 36539736
- [Derived] Kim NY, Park JH, Park J, Kwak N, Choi SM, Park YS, Lee CH, Cho J. Effect of Chlorhexidine Mouthrinse on Prevention of Microbial Contamination during EBUS-TBNA: A Study Protocol for a Randomized Controlled Trial. Tuberc Respir Dis (Seoul). 2021 Oct;84(4):291-298. doi: 10.4046/trd.2021.0058. Epub 2021 Jun 24. PMID 34162198